CLINICAL TRIAL: NCT04830514
Title: Maximizing the Dietary Pattern of Older Adults: the Effects of Protein Intake on Protein Kinetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 262424
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Results first posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2022-10

CONDITIONS: Sarcopenia
Keywords: muscle loss; protein; animal-based protein
MeSH Terms: conditions — Sarcopenia; Muscular Atrophy | interventions — Nutrition Surveys

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Recommended dietary allowance (RDA) for protein (Experimental): (RDA; 0.8g/kg/day) Protein intakes will be structured within two meals per day. A 2-day dietary lead-in will precede each dietary intervention. Study duration per subject will last about two weeks.
  Interventions: Other: Recommended Dietary Allowance of Protein
- Habitual protein intake consistent with population level norms (Experimental): (NHANES; 1.0g/kg/day) Protein intakes will be structured within two meals per day. A 2-day dietary lead-in will precede each dietary intervention. Study duration per subject will last about two weeks.
  Interventions: Other: Habitual protein intake
- Optimal protein intake (OPI) (Experimental): (OPI; 1.5g/kg/day) Protein intakes will be structured within two meals per day. A 2-day dietary lead-in will precede each dietary intervention. Study duration per subject will last about two weeks.
  Interventions: Other: Optimal Protein Intake

INTERVENTIONS:
Other: Recommended Dietary Allowance of Protein — 0.8 g/kg/day protein intake
  Other Names: RDA
  Arms: Recommended dietary allowance (RDA) for protein
Other: Habitual protein intake — 1.0 g/kg/day protein intake
  Other Names: NHANES
  Arms: Habitual protein intake consistent with population level norms
Other: Optimal Protein Intake — 1.5 g/kg/day protein intake
  Other Names: OPI
  Arms: Optimal protein intake (OPI)

SUMMARY:
A randomized study to demonstrate how animal-based protein-rich food sources can be used by older adults to increase protein intake within pre-existing dietary patterns.

DETAILED DESCRIPTION:
Current dietary patterns of older Americans will be augmented by readily available quality protein sources. Investigators will observe the effects of recommended and common protein intakes on the maintenance of whole-body protein balance and potential for muscle protein anabolism.

3 groups of 10 older subjects will be studied during daily protein intakes. Study duration per subject will be about 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≤ 35 kg/m2
* Capable of providing informed consent
* COVID-19 negative and/or asymptomatic

Exclusion Criteria:

* Subject who does not/will not eat animal protein sources.
* Body mass index > 35.
* History of chemotherapy or radiation therapy for cancer in the 6 months prior to enrollment.
* Use of insulin to control blood sugar level.
* Currently receiving androgen (e.g., testosterone) or anabolic (e.g., GH, IGF-I) therapy.
* Currently using prescription blood thinning medications.
* Unable or unwilling to suspend aspirin use for 7 days prior to Visit 3.
* Unwilling to avoid using protein or amino-acid supplements during participation.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arny A Ferrando, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Church DD, Hirsch KR, Kviatkovsky SA, Matthews JJ, Henderson RA, Azhar G, Wolfe RR, Ferrando AA. Effect of 3 Different Daily Protein Intakes in a 2-Meal Eating Pattern on Protein Turnover in Middle Age and Older Adults: A Randomized Controlled Trial. J Nutr. 2025 May;155(5):1364-1372. doi: 10.1016/j.tjnut.2024.12.025. Epub 2024 Dec 28. PMID 39736329

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Recommended Dietary Allowance (RDA) for Protein | Habitual Protein Intake Consistent With Population Level Norms | Optimal Protein Intake (OPI)
Started | 18 | 14 | 12
Completed | 10 | 11 | 9
Not Completed | 8 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Recommended Dietary Allowance (RDA) for Protein | Habitual Protein Intake Consistent With Population Level Norms | Optimal Protein Intake (OPI) | Total
Number analyzed (Participants) | 10 | 11 | 9 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 9 | 24
  >=65 years | 3 | 3 | 0 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 6 | 17
  Male | 5 | 5 | 3 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 11 | 9 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 9 | 10 | 7 | 26
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 9 | 30

OUTCOME MEASURES:

1. Primary Outcome: Whole Body Protein Turnover
Description: Isotope Tracer
Time Frame: 24 hour
Measure: Mean (Standard Deviation); unit: g/kg lean body mass/day
Arm/Group | Recommended Dietary Allowance (RDA) for Protein | Habitual Protein Intake Consistent With Population Level Norms | Optimal Protein Intake (OPI)
Number analyzed (Participants) | 10 | 11 | 9
g/kg lean body mass/day | -0.16 (0.08) | -0.17 (0.11) | 0.48 (0.11)

ADVERSE EVENTS:
Time Frame: Starting with enrollment and ending with completion of last study visit; in most cases within 30 days.
Arm/Group | Recommended Dietary Allowance (RDA) for Protein | Habitual Protein Intake Consistent With Population Level Norms | Optimal Protein Intake (OPI)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 6/18 | 3/14 | 5/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recommended Dietary Allowance (RDA) for Protein (N=18) | Habitual Protein Intake Consistent With Population Level Norms (N=14) | Optimal Protein Intake (OPI) (N=12)
Laceration from fall (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Subject fell and hit their head on the edge of a nearby table, causing a deep scalp laceration.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recommended Dietary Allowance (RDA) for Protein (N=18) | Habitual Protein Intake Consistent With Population Level Norms (N=14) | Optimal Protein Intake (OPI) (N=12)
Laceration from fall (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Ear and labyrinth disorders) | 5 (5) | 2 (2) | 5 (5)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
GI illness with reflux (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/14/NCT04830514/Prot_SAP_000.pdf